CLINICAL TRIAL: NCT00337883
Title: A Phase II, Multicenter, Open-Label Trial of the Safety and Efficacy of Tarceva (Erlotinib Hydrochloride) in Patients With First Relapse of Grade IV Glioma (Glioblastoma Multiforme)
Brief Title: A Study of the Safety and Efficacy of Tarceva in Patients With First Relapse of Grade IV Glioma (Glioblastoma Multiforme)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: OSI2691g; NCT00090883 (obsolete NCT alias)
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Glioblastoma
Keywords: Glioblastoma Multiforme; glioma; Grade IV glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib HCl (OSI-774)

SUMMARY:
This is a Phase II, open-label, multicenter trial of single-agent treatment with Tarceva in patients with histologically confirmed GBM in first relapse. This study seeks to estimate the objective response rate and will investigate whether response rate is related to EGFR amplification status.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >= 18 years
* Histologically confirmed GBM in first relapse
* Disease progression in those patients following prior implantation with Gliadel(R) wafer(s) (polifeprosan 20 with carmustine implant) must be confirmed by biopsy. Prior therapy with Gliadel(R) is allowed only as a component of primary surgery. Patients with Gliadel(R) implants after a secondary resection are not eligible.
* Radiographic evidence of disease progression, as assessed by the investigator, on magnetic resonance imaging (MRI) or CT scan
* Bi-dimensionally measurable disease with a minimum measurement of 1 cm on MRI or CT scan performed within 14 days prior to study entry
* Prior radiotherapy
* Availability of tissue to allow central confirmation of GBM diagnosis (all original slides are preferred)
* Availability of paraffin blocks or slides to allow determination of EGFR amplification status
* Recovery from the toxic effects of a prior therapy, including 4 weeks from prior cytotoxic agents (except 6 weeks from prior nitrosoureas, 3 weeks from prior procarbazine administration, 2 weeks from prior vincristine, or 3 weeks from irinotecan [CPT-11] when given on a weekly schedule), 4 weeks from any prior investigational agent, and 1 week from prior non-cytotoxic agents (e.g., interferon, tamoxifen, thalidomide, 13-cis-retinoic acid, etc.)
* If receiving corticosteroids, patients must be on a stable, non-increasing dose of corticosteroids for >= 2 weeks prior to baseline MRI scan
* ECOG performance status of 0 or 1
* Life expectancy > 12 weeks
* Use of an effective means of contraception in males and in females of childbearing potential
* Ability to comply with study and follow-up procedures If the decision is made at the end of Stage 1 to enroll patients with tumors known to be positive for EGFR amplification, the following additional inclusion criteria will be applied: Confirmation of diagnosis; Confirmation of positive EGFR amplification status

Exclusion Criteria:

* Prior treatment with Gleevec (e.g., imatinib mesylate) or agents directed at EGFR (e.g., Iressa)
* Prior treatment with Gliadel(R) following second (salvage or debulking) therapy
* History of any other malignancy within 5 years (except non-melanoma skin cancer or carcinoma in situ of the cervix)
* More than one prior chemotherapy regimen
* ANC < 1500/uL
* Platelets < 100,000/uL
* Total bilirubin > 1.6 mg/dL
* AST/ALT >= 2.5 x upper limit of normal (ULN)
* Creatinine > 1.5 x ULN
* Pregnant or nursing females
* Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to study entry, or serious cardiac arrhythmia requiring medication
* Major surgical procedure 2 weeks prior to study entry or anticipation of need for major surgical procedure during the course of the study
* Inability to take oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2003-07; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Klencke, M.D., Study Director — Genentech, Inc.